CLINICAL TRIAL: NCT00426452
Title: A Phase IB, Open Label, Single Center, Drug-drug Interaction Study of Oral 1250 mg of PTK787/ZK 222584 Administered Under Fasting and Fed Conditions With a Proton-pump Inhibitor (Omeprazole) in Healthy Sterile or Postmenopausal Female Volunteers
Brief Title: A Drug-drug Interaction Study of Oral 1250 mg of Vatalinib Administered Under Fasting and Fed Conditions With a Proton-pump Inhibitor in Healthy Sterile or Postmenopausal Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Bayer (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPTK787A2121
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Vascular endothelial growth factor receptor (VEGF-R) tyrosine kinase inhibitor; Vatalinib; Proton-pump inhibitors; Omeprazole; Healthy Postmenopausal Female Volunteers
MeSH Terms: interventions — vatalanib

INTERVENTIONS:
Drug: Vatalinib

SUMMARY:
This study will determine the effect of acidic drugs such as proton-pump inhibitors on the pharmacokinetics of Vatalinib under fasting and fed conditions.

ELIGIBILITY:
Inclusion criteria

* Healthy female
* Surgically sterile or post-menopausal
* At least a weight of 50 kg and have a body mass index (BMI) ≤33.0
* Non-smokers or those who smoke 25 cigarettes or less per day Exclusion criteria
* Use of certain prescription and over the counter drugs
* Having received an investigational drug within 30 days prior to dosing
* Donation of plasma or donation or loss of whole blood prior to administration of the study medication
* Any clinically significant laboratory tests
* Abnormal cardiac function
* A positive test for HIV, Hepatitis B or C
* A positive alcohol test or drug test
* Known allergy to Vatalinib or Omeprazole
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism and excretion or drugs.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 35 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-07

PRIMARY OUTCOMES:
Assess the effect of multiple doses of a proton-pump inhibitor on the pharmacokinetics of a single dose of Vatalinib under fasting and fed conditions.

SECONDARY OUTCOMES:
Safety of a single dose of Vatalinib before and after a proton-pump inhibitor under fasting and fed conditions as assessed by adverse events, laboratory values, electrocardiograms, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis